CLINICAL TRIAL: NCT03043573
Title: Problem Adaptation Therapy for Mild Cognitive Impairment and Depression
Acronym: PATH-MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Johns Hopkins University (Other); Montefiore Medical Center (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1603017114; 1R01AG050514 (NIH)
Record Dates: First submitted 2017-01-27; First posted 2017-02-06 (Estimated); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Cognitive Impairment; Depression
MeSH Terms: conditions — Cognitive Dysfunction; Depression | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PATH-MCI (Experimental): Problem Adaptation Therapy for Mild Cognitively Impaired Adults (PATH-MCI) differs from standard of care psychotherapy by offering a combination of emotion regulation techniques with the provision of environmental adaptation tools (notes, checklists, calendars, etc.), the use of the WellPATH app, and the participation of a willing and available caregiver.
  Interventions: Behavioral: PATH-MCI
- Supportive Therapy (Active Comparator): Supportive Therapy focuses on: 1. Facilitating expression of affect; 2. Conveying to the patient that he or she is understood; 3. Offering empathy; and 4. Highlighting positive experiences. The ST manual aims to standardize nonspecific therapeutic factors.
  Interventions: Behavioral: Supportive Therapy

INTERVENTIONS:
Behavioral: PATH-MCI — Problem Adaptation Therapy for Mild Cognitively Impaired Adults (PATH-MCI) differs from standard of care psychotherapy by offering a combination of emotion regulation techniques with the provision of environmental adaptation tools (notes, checklists, calendars, etc.), the use of the WellPATH app, and the participation of a willing and available caregiver.
  Arms: PATH-MCI
Behavioral: Supportive Therapy — ST focuses on: 1. facilitating expression of affect; 2. conveying to the patient that he or she is understood; 3. offering empathy; and 4. highlighting positive experiences. The ST manual aims to standardize nonspecific therapeutic factors.
  Other Names: ST
  Arms: Supportive Therapy

SUMMARY:
The present collaborative R01 study, between Cornell and Johns Hopkins, aims to compare Problem Adaptation Therapy for Mild Cognitively Impaired Older Adults (PATH-MCI) vs. Supportive Therapy for Cognitively Impaired Older Adults (ST-CI) in improving cognitive, affective, and functioning outcomes.

DETAILED DESCRIPTION:
The present collaborative R01 study, between Cornell and Johns Hopkins, aims to compare Problem Adaptation Therapy for Mild Cognitively Impaired Older Adults (PATH-MCI) vs. Supportive Therapy for Cognitively Impaired Older Adults (ST-CI) in improving cognitive, affective and functioning outcomes. Psychotherapy, also known as talking therapy, is the use of psychological methods to help a person change and overcome problems in desired ways. PATH-MCI differs from standard of care psychotherapy by offering a combination of emotion regulation techniques with the provision of environmental adaptation tools (notes, checklists, calendars, etc.), the use of the WellPATH app, and the participation of a willing and available caregiver. Supportive Therapy incorporates standard of care approaches by using non-specific techniques to provide a supportive environment and help patients to express their feelings & focus on their strengths and abilities.

The investigators plan to randomize 80 treatment subjects, older adults (40 at Cornell and 40 at Johns Hopkins) with MCI-depression. 80 study partners may also be potentially recruited. Both sites have shown feasibility of recruitment, randomization, retention, and assessment procedures for patients with MCI. Cornell has shown evidence of administration of PATH in this population. Certified mental health clinicians in PATH-MCI and ST-CI will administer 15 in-office sessions in six months.

The investigators propose to compare the effects of 15 sessions (12 weekly in first 12 weeks and 3 monthly booster sessions afterwards) of PATH-MCI vs. ST-CI in 80 older adults (treatment subjects) with MCI-depression. Research assistants, unaware of study hypotheses and participant randomization status, will perform research assessments at baseline and at 6 (no cognitive measures), 12, 24, 36 (no cognitive measures) and 52 weeks after randomization.

There will also be optional blood draws at study entry, 12, and 52 weeks. The purpose of the blood draws is to better understand whether response to psychotherapy treatment is affected by genes, by inflammation, or by the possible memory factor called BDNF (brain-derived neurotrophic factor). Also, all therapy sessions will be audiotaped (if the patient consents) and Dr. Shermer (a clinician outside of the Weill Cornell Institute of Geriatric Psychiatry) will evaluate randomly selected sessions and rate the therapists' adherence and competence based on the PATH-MCI and ST Adherence Scales

The study partner will provide information about the treatment subject and participate in treatment if agreed by the treatment subject. To explore the effects of PATH-MCI on the study partner, the investigators will collect the following data from the study partner: demographic, burden (Short Zarit Burden interview), and treatment satisfaction (Client Satisfaction Questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Amnestic MCI as defined by Albert et al
* Montgomery Asberg Depression Rating Scale (MADRS) greater than 7 and MADRS total less than 30
* Participants will be off antidepressants, cholinesterase inhibitors or memantine, or on a stable dosage for at least 12 weeks without any medical recommendation to adjust dosage in next 3 months (during treatment)
* Clinical Dementia Rating (CDR) = 0.5 at screening
* Subjects will have capacity to consent

Exclusion Criteria:

* Deemed to have a significant suicide risk as assessed by site PI and clinical team
* Deemed too unstable medically or neurologically to safely enroll in a research trial
* Deemed too psychiatrically unstable to safely enroll in randomized trial of psychotherapy. Requiring psychiatric hospitalization at baseline for safety.
* Current involvement in psychotherapy
* Lack of English fluency

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Kiosses, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Weill Cornell Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Weill Cornell Institute of Geriatric Psychiatry, Weill Cornell Medicine, White Plains, New York

IPD SHARING:
Plan to Share IPD: Yes
Data will be available as per NIH's data sharing policy.
Time Frame: Data will be available as per NIH's data sharing policy.
Access Criteria: Access criteria is determined by NIH and can be requested by applying online.
URL: https://nda.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PATH-MCI | Supportive Therapy
Started | 39 | 41
Completed | 36 | 29
Not Completed | 3 | 12
Not completed — Lost to Follow-up | 3 | 3
Not completed — Physician Decision | 0 | 5
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PATH-MCI | Supportive Therapy | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.87 (7.82) | 73.56 (7.42) | 73.71 (7.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 17 | 21 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 38 | 37 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 34 | 33 | 67
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Cognition Assessed by RBANS
Description: Global cognition will be assessed by the Repeatable Battery for the Assessment of Neuropsychological Status Total Score (RBANS). The total score represents the simple sum of the five cognitive domain index scores (Immediate Memory, Visuospatial/Constructional, Language, Attention, and Delayed Memory). Total raw scores are converted based on the subjects age and a RBANS scoring manual. Higher scores indicate better functionality. The total scores range from 200 to 800.
Time Frame: Baseline, 12, 24, and 52 Weeks
Population: The study was affected by the pandemic and by the inability of certain participants to complete assessment measures during the study. Therefore, there is a discrepancy between the numbers of randomized and the numbers of analyzed participants at different time points.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | PATH-MCI | Supportive Therapy
Number analyzed (Participants) | 38 | 39
Score on a Scale
  Baseline Totals | 434.66 (68.96) | 435.36 (68.27)
  Week 12 Totals: number analyzed (Participants) | 37 | 27
  Week 12 Totals | 438.46 (70.27) | 436 (67.51)
  Week 24 Totals: number analyzed (Participants) | 35 | 24
  Week 24 Totals | 448.57 (71.78) | 449.08 (64.75)
  Week 52 Totals: number analyzed (Participants) | 26 | 21
  Week 52 Totals | 435 (111.04) | 419.33 (101.93)
Statistical Analysis 1: Comparison: PATH-MCI vs Supportive Therapy; Baseline; Test type: Superiority; p = 0.9644, t-test, 2 sided; Mean Difference (Final Values) = -0.7011, 95% CI 2-sided [-31.8605 to 30.4583]
Statistical Analysis 2: Comparison: PATH-MCI vs Supportive Therapy; Week 12; Test type: Superiority; p = 0.8880, t-test, 2 sided; Mean Difference (Final Values) = 2.4595, 95% CI 2-sided [-32.3472 to 37.2661]
Statistical Analysis 3: Comparison: PATH-MCI vs Supportive Therapy; Week 24; Test type: Superiority; p = 0.9773, t-test, 2 sided; Mean Difference (Final Values) = -0.5119, 95% CI 2-sided [-36.5024 to 35.4785]
Statistical Analysis 4: Comparison: PATH-MCI vs Supportive Therapy; Week 52; Test type: Superiority; p = 0.6173, t-test, 1 sided; Mean Difference (Final Values) = 15.6667, 95% CI 2-sided [-47.0598 to 78.3931]

2. Secondary Outcome: Change in Disability Function Assessed With WHODAS-II
Description: The 12-item WHODAS-II (World Health Organization Disability Assessment Schedule) assesses functional impairment across six domains of daily living. Each item is scored on a 5-point Likert scale ranging from 0 (No difficulty), 1 (Mild Difficulty), 2 (Moderate Difficulty), 3 (Severe Difficulty) and 4 (Extreme difficulty or cannot do). Each individual item has a minimum score of 0 and a maximum of 4. The total raw score is computed by summing all 12 items, resulting in a possible score range of 0 to 48. Higher score reflect greater functional impairment. Lower scores indicate better functional status and less reported difficulty with daily activities.
Time Frame: Baseline, 6, 12, 24, 36, and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | PATH-MCI | Supportive Therapy
Number analyzed (Participants) | 38 | 39
Score on a Scale
  Baseline Totals | 12.08 (7.74) | 10.95 (8.57)
  Week 6 Totals: number analyzed (Participants) | 37 | 34
  Week 6 Totals | 12.43 (8.72) | 9.47 (7.16)
  Week 12 Totals: number analyzed (Participants) | 37 | 31
  Week 12 Totals | 10.68 (7.55) | 9.58 (8.17)
  Week 24 Totals: number analyzed (Participants) | 35 | 30
  Week 24 Totals | 8.51 (8.01) | 10.07 (7.97)
  Week 36 Totals: number analyzed (Participants) | 34 | 26
  Week 36 Totals | 9.97 (8.45) | 9.08 (8.19)
  Week 52 Totals: number analyzed (Participants) | 28 | 25
  Week 52 Totals | 11.79 (8.67) | 8.84 (6.36)
Statistical Analysis 1: Comparison: PATH-MCI vs Supportive Therapy; Baseline; Test type: Superiority; p = 0.5454, t-test, 2 sided; Mean Difference (Final Values) = 1.1302, 95% CI 2-sided [-2.5767 to 4.8371]
Statistical Analysis 2: Comparison: PATH-MCI vs Supportive Therapy; Week 6; Test type: Superiority; p = 0.1212, t-test, 2 sided; Mean Difference (Final Values) = 2.9618, 95% CI 2-sided [-0.8038 to 6.7275]
Statistical Analysis 3: Comparison: PATH-MCI vs Supportive Therapy; Week 12; Test type: Superiority; p = 0.5710, t-test, 2 sided; Mean Difference (Final Values) = 1.0950, 95% CI 2-sided [-2.7476 to 4.9377]
Statistical Analysis 4: Comparison: PATH-MCI vs Supportive Therapy; Week 24; Test type: Superiority; p = 0.4377, t-test, 2 sided; Mean Difference (Final Values) = -1.5524, 95% CI 2-sided [-5.5256 to 2.4209]
Statistical Analysis 5: Comparison: PATH-MCI vs Supportive Therapy; Week 36; Test type: Superiority; p = 0.6813, t-test, 2 sided; Mean Difference (Final Values) = 0.8937, 95% CI 2-sided [-3.4439 to 5.2312]
Statistical Analysis 6: Comparison: PATH-MCI vs Supportive Therapy; Test type: Superiority; p = 0.1620, t-test, 2 sided; Mean Difference (Final Values) = 2.9457, 95% CI 2-sided [-1.2234 to 7.1148]

3. Secondary Outcome: Change in Depression Assessed by MADRS
Description: Depression assessed by Montgomery Asberg Depression Rating Scale (MADRS) Total Score. The MADRS is a 10 item questionnaire assessing severity of depression by scoring participants on mood, anxiety, sleep, concentration, appetite, and suicidal thoughts. The lowest score is 0, no depression symptoms, and the highest possible score is 60, severe depression symptoms.
Time Frame: Baseline, 6, 12, 24, 36, and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | PATH-MCI | Supportive Therapy
Number analyzed (Participants) | 37 | 39
Score on a Scale
  Baseline Totals | 16.62 (5.8) | 16.59 (6.01)
  Week 6 Totals: number analyzed (Participants) | 37 | 34
  Week 6 Totals | 14.97 (8.57) | 15.03 (5.47)
  Week 12 Totals: number analyzed (Participants) | 36 | 30
  Week 12 Totals | 13.53 (6.81) | 12.47 (6.38)
  Week 24 Totals: number analyzed (Participants) | 36 | 30
  Week 24 Totals | 10.67 (6.61) | 12.67 (5.85)
  Week 36 Totals: number analyzed (Participants) | 34 | 26
  Week 36 Totals | 12.32 (6.4) | 11.96 (6.76)
  Week 52 Totals: number analyzed (Participants) | 27 | 25
  Week 52 Totals | 12.67 (6.17) | 11.4 (6.40)
Statistical Analysis 1: Comparison: PATH-MCI vs Supportive Therapy; Baseline; Test type: Superiority; p = 0.9813, t-test, 2 sided; Mean Difference (Final Values) = 0.0319, 95% CI 2-sided [-2.6668 to 2.7305]
Statistical Analysis 2: Comparison: PATH-MCI vs Supportive Therapy; Week 6; Test type: Superiority; p = 0.9735, t-test, 2 sided; Mean Difference (Final Values) = -0.0564, 95% CI 2-sided [-3.4397 to 3.3268]
Statistical Analysis 3: Comparison: PATH-MCI vs Supportive Therapy; Test type: Superiority — Week 12; p = 0.5164, t-test, 2 sided; Mean Difference (Final Values) = 1.0611, 95% CI 2-sided [-2.1885 to 4.3107]
Statistical Analysis 4: Comparison: PATH-MCI vs Supportive Therapy; Week 24; Test type: Superiority; p = 0.1970, t-test, 2 sided; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-5.0651 to 1.0651]
Statistical Analysis 5: Comparison: PATH-MCI vs Supportive Therapy; Week 36; Test type: Superiority; p = 0.8342, t-test, 2 sided; Mean Difference (Net) = 0.3620, 95% CI 2-sided [-3.0907 to 3.8146]
Statistical Analysis 6: Comparison: PATH-MCI vs Supportive Therapy; Week 52; Test type: Superiority; p = 0.4717, t-test, 2 sided; Mean Difference (Final Values) = 1.2667, 95% CI 2-sided [-2.2424 to 4.7758]

4. Secondary Outcome: Change in Episodic Memory Assessed by Delayed Recall Subscale of RBANS
Description: The Delayed Recall subscale of the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) assesses memory function across multiple tasks. It includes the following components: List Recall Total Score (range: 0-10), List Recognition Total Score (range: 0-20), Story Recall Total Score (range: 0-12), and Figure Recall Total Score (range: 0-20). The raw scores from these four components are summed to yield a Delayed Memory Index raw total score ranging from 0 to 62, with higher scores indicating better memory performance.
  To facilitate standardized interpretation, raw total scores are converted to age-adjusted Index Scores using normative data provided in the RBANS manual. These Index Scores have a mean of 100 and a standard deviation of 15, and are normed by decade (e.g., 60-69, 70-79, 80-89). Higher Index Scores reflect better memory functioning relative to age-matched peers.
Time Frame: Baseline, 12, 24, and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | PATH-MCI | Supportive Therapy
Number analyzed (Participants) | 38 | 39
Score on a Scale
  Baseline Totals | 76.66 (20.18) | 79.59 (18.92)
  Week 12 Totals: number analyzed (Participants) | 37 | 27
  Week 12 Totals | 77.81 (22.36) | 81.78 (22.12)
  Week 24 Totals: number analyzed (Participants) | 35 | 24
  Week 24 Totals | 81.89 (21.89) | 87.04 (20.40)
  Week 52 Totals: number analyzed (Participants) | 24 | 20
  Week 52 Totals | 84.71 (22.91) | 83.60 (23.66)
Statistical Analysis 1: Comparison: PATH-MCI vs Supportive Therapy; Baseline; Test type: Superiority; p = 0.5130, t-test, 2 sided; Mean Difference (Final Values) = -2.9318, 95% CI 2-sided [-11.8176 to 5.9539]
Statistical Analysis 2: Comparison: PATH-MCI vs Supportive Therapy; Week 12; Test type: Superiority; p = 0.4835, t-test, 2 sided; Mean Difference (Final Values) = 0.4835, 95% CI 2-sided [-15.2306 to 7.2967]
Statistical Analysis 3: Comparison: PATH-MCI vs Supportive Therapy; Week 24; Test type: Superiority; p = 0.3590, t-test, 2 sided; Mean Difference (Final Values) = -5.1560, 95% CI 2-sided [-16.3357 to 6.0238]
Statistical Analysis 4: Comparison: PATH-MCI vs Supportive Therapy; Week 52; Test type: Superiority; p = 0.8760, t-test, 2 sided; Mean Difference (Final Values) = 1.1083, 95% CI 2-sided [-13.1598 to 15.3765]

5. Secondary Outcome: Change in Executive Function Assessed by Trail Making Test
Description: Trail Making Test is a neuropsychological assessment where raw scores are converted into a scaled score range from 1 to 25. Participants with scores between 1 - 8 have impaired performance; Mid range scores typically fall between 10 - 16, and subjects who fair the best on this measure have scores ranging from 20 - 25.
Time Frame: Baseline, 12, 24, and 52 Weeks
Population: The study was affected by the pandemic and by the inability of certain participants to complete assessment measures during the study. Therefore, there is a discrepancy between the numbers of randomized and the numbers of analyzed participants at different time points. Trails A consists of the numbers being connected in sequence. Trails B alternate between numbers and letters.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | PATH-MCI | Supportive Therapy
Number analyzed (Participants) | 33 | 30
Score on a Scale
  Baseline Totals (Trails A): number analyzed (Participants) | 33 | 29
  Baseline Totals (Trails A) | 24.94 (0.35) | 25 (0.00)
  Week 12 Totals (Trails A): number analyzed (Participants) | 31 | 18
  Week 12 Totals (Trails A) | 24.19 (4.13) | 24.89 (0.47)
  Week 24 Totals (Trails A): number analyzed (Participants) | 28 | 16
  Week 24 Totals (Trails A) | 25 (0.00) | 25 (0.00)
  Week 52 Totals (Trails A): number analyzed (Participants) | 14 | 10
  Week 52 Totals (Trails A) | 25 (0.00) | 25 (0.00)
  Baseline Totals (Trails B): number analyzed (Participants) | 32 | 30
  Baseline Totals (Trails B) | 23.63 (5.16) | 22.63 (6.36)
  Week 12 Totals (Trails B): number analyzed (Participants) | 31 | 17
  Week 12 Totals (Trails B) | 22.65 (5.96) | 24.71 (0.85)
  Week 24 Totals (Trails B): number analyzed (Participants) | 28 | 16
  Week 24 Totals (Trails B) | 24.11 (3.33) | 25 (0.00)
  Week 52 Totals (Trails B): number analyzed (Participants) | 14 | 10
  Week 52 Totals (Trails B) | 23.57 (4.13) | 25 (0.00)
Statistical Analysis 1: Comparison: PATH-MCI vs Supportive Therapy; Trails A Baseline; Test type: Superiority; p = 0.3248, t-test, 2 sided; Mean Difference (Final Values) = -0.0606, 95% CI 2-sided [-0.1841 to 0.0628]
Statistical Analysis 2: Comparison: PATH-MCI vs Supportive Therapy; Trails A - Week 12; Test type: Superiority; p = 0.3615, t-test, 2 sided; Mean Difference (Final Values) = -0.6953, 95% CI 2-sided [-2.2261 to 0.8354]
Statistical Analysis 3: Comparison: PATH-MCI vs Supportive Therapy; Trails B - Baseline; Test type: Superiority; p = 0.5046, t-test, 2 sided; Mean Difference (Final Values) = 0.9917, 95% CI 2-sided [-1.9664 to 3.9498]
Statistical Analysis 4: Comparison: PATH-MCI vs Supportive Therapy; Trails B - Week 12; Test type: Superiority; p = 0.0679, t-test, 2 sided; Mean Difference (Final Values) = -2.0607, 95% CI 2-sided [-4.2821 to 0.1607]
Statistical Analysis 5: Comparison: PATH-MCI vs Supportive Therapy; Trails B - Week 24; Test type: Superiority; p = 0.1669, t-test, 2 sided; Mean Difference (Final Values) = -0.8929, 95% CI 2-sided [-2.1825 to 0.3968]
Statistical Analysis 6: Comparison: PATH-MCI vs Supportive Therapy; Trails B - Week 52; Test type: Superiority; p = 0.2178, t-test, 2 sided; Mean Difference (Final Values) = -1.4286, 95% CI 2-sided [-3.8115 to 0.9543]

6. Other Pre Specified Outcome: Change in Stress Reduction Assessed by Perceived Stress Scale
Description: Perceived Stress Scale s the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. The 10-item measure has 4 choice options; (0=Never, 1=Almost Never, 2=Sometimes, 3=Fairly Often, 4=Often). 4 items are reversed scored and the total score is summed across all items ranging from 0 to 40. Lower scores are better and indicate less stress.
Time Frame: Baseline, 6, 12, 24, 36, and 52 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | PATH-MCI | Supportive Therapy
Number analyzed (Participants) | 38 | 39
Score on a Scale
  Baseline Totals | 19.76 (6.81) | 18.21 (6.07)
  Week 6 Totals: number analyzed (Participants) | 37 | 34
  Week 6 Totals | 18.35 (7.45) | 16.65 (5.90)
  Week 12 Totals: number analyzed (Participants) | 36 | 30
  Week 12 Totals | 17.25 (7.48) | 16.33 (6.31)
  Week 24 Totals: number analyzed (Participants) | 35 | 30
  Week 24 Totals | 16.34 (8.33) | 17.37 (7.88)
  Week 36 Totals: number analyzed (Participants) | 34 | 26
  Week 36 Totals | 16.24 (7.96) | 14.31 (7.26)
  Week 52 Totals: number analyzed (Participants) | 27 | 24
  Week 52 Totals | 17.07 (7.85) | 15.00 (6.06)
Statistical Analysis 1: Comparison: PATH-MCI vs Supportive Therapy; Baseline; Test type: Superiority; p = 0.2932, t-test, 2 sided; Mean Difference (Final Values) = 1.5580, 95% CI 2-sided [-1.3747 to 4.4908]
Statistical Analysis 2: Comparison: PATH-MCI vs Supportive Therapy; Week 6; Test type: Superiority; p = 0.2871, t-test, 2 sided; Mean Difference (Final Values) = 1.7043, 95% CI 2-sided [-1.4659 to 4.8744]
Statistical Analysis 3: Comparison: PATH-MCI vs Supportive Therapy; Week 12; Test type: Superiority; p = 0.5910, t-test, 2 sided; Mean Difference (Final Values) = 0.9167, 95% CI 2-sided [-2.4737 to 4.3070]
Statistical Analysis 4: Comparison: PATH-MCI vs Supportive Therapy; Test type: Superiority; p = 0.6128, t-test, 2 sided; Mean Difference (Final Values) = -1.0238, 95% CI 2-sided [-5.0469 to 2.9993]
Statistical Analysis 5: Comparison: PATH-MCI vs Supportive Therapy; Week 36; Test type: Superiority; p = 0.3326, t-test, 2 sided; Mean Difference (Final Values) = 1.9276, 95% CI 2-sided [-2.0231 to 5.8783]
Statistical Analysis 6: Comparison: PATH-MCI vs Supportive Therapy; Week 52; Test type: Superiority; p = 0.2935, t-test, 2 sided; Mean Difference (Final Values) = 2.0741, 95% CI 2-sided [-1.8522 to 6.0004]

ADVERSE EVENTS:
Time Frame: 52 Weeks
Arm/Group | PATH-MCI | Supportive Therapy
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/41
Serious Adverse Events (participants affected / at risk) | 5/39 | 1/41
Other Adverse Events (participants affected / at risk) | 4/39 | 6/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PATH-MCI (N=39) | Supportive Therapy (N=41)
Major Depressive Episode (Psychiatric disorders) | 1 (1) | 0 (0)
Masectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Breast Reconstruction (Surgical and medical procedures) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PATH-MCI (N=39) | Supportive Therapy (N=41)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin Biopsy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Retinal Detachment (Endocrine disorders) | 0 (0) | 1 (1)
Laminectomy and discectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Skin Lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT03043573/Prot_000.pdf
  • Informed Consent Form (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT03043573/ICF_001.pdf